CLINICAL TRIAL: NCT05343741
Title: Practice-Based Evidence in Ecuador: Routine Outcome Monitoring in Psychotherapy for Common Mental Health Problems
Brief Title: Practice-Based Evidence in Psychotherapy in Ecuador
Status: Active, not recruiting | Type: Observational
Sponsor: Universidad de las Americas - Quito (Other)
Responsible Party: Principal Investigator, Jorge Valdiviezo Oña, Prof., Universidad de las Americas - Quito
Other Study IDs: 20211202_jvaldiviezo
Record Dates: First submitted 2022-03-31; First posted 2022-04-25 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Psychological Distress
Keywords: practice-based evidence; routine outcome monitoring; psychotherapy; change; outcome; psychological distress
MeSH Terms: interventions — Psychosocial Intervention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Helpseeking Ecuadorian adult and adolescent clients: The participants will be adolescent (11-17 years) and adult (>18 years) clients presenting with common non-severe mental health problems who seek mental health services at the Centro de Psicología Aplicada. The CPA is an outpatient psychological service where students of the last semesters of the Clinical Psychology degree develop and practice their psychological care skills as co-therapists of professional clinical psychologists.
  Interventions: Other: Psychological Intervention

INTERVENTIONS:
Other: Psychological Intervention — The CPA provides outpatient psychological services to individuals: children, adolescents and adults, couples and families. At the CPA, care is carried out through the co-therapy model, which involves the participation of a professional clinical psychologist and a trainee. Psychotherapists with diverse theoretical and clinical backgrounds (mainly psychodynamic, cognitive, systemic and integrative), but a common constructivist approach, work in the center. The following elements are transversal in their practice: therapeutic alliance, healing environment, and a collaborative procedure between the client, the psychotherapist and the trainee co-therapist.

SUMMARY:
This is a naturalistic study implementing a routine outcome monitoring system to track clients' change and outcomes at the Centro de Psicología Aplicada (CPA) of the Universidad de Las Américas in Quito, Ecuador

DETAILED DESCRIPTION:
This is an exploratory and descriptive naturalistic longitudinal project. The general objective of this study is to systematically examine the progress and outcomes of psychological interventions provided at the Centro de Psicología Aplicada (CPA) of the Universidad de Las Américas by routinely monitoring outcomes through an standardized system.

Characteristics of the participants and the received interventions will be recorded through the use of assessment forms filled by therapists before and after therapy, and clients will complete outcome measures on psychological distress, life satisfaction, ambivalence in psychotherapy, family functioning, therapeutic alliance, and satisfaction with the treatment received.

This is the first project in Ecuador to propose a system for routine outcome monitoring in psychotherapy. It could contribute to develop normative trajectories of change and expected recovery curves in the future and to improve the quality of psychological treatments.

ELIGIBILITY:
Inclusion Criteria:

* Be 11 years of age or older.
* Have sufficient ability to communicate in Spanish.
* Undergo psychological treatment at the CPA.

Exclusion Criteria:

* Present substantial cognitive deficits that do not allow the development of the evaluation.

Ages: 11 Years to 100 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Helpseeking clients undergoing treatment at the Centro de Psicología Aplicada of the Universidad de Las Américas
Sampling Method: Non-Probability Sample
Enrollment: 340 (Estimated)
Dates: Start 2022-10-17 (Actual); Primary Completion 2025-07-20 (Actual); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in Clinical Outcomes in Routine Evaluation-Outcome Measure (CORE-OM) | CORE-OM is administered to adult clients at baseline and immediately after treatment completion
  The CORE-OM (Evans et al., 2002) is a 34-item self-report instrument designed for use in heterogeneous services and based on a pan-theoretic core of psychological distress, including subjective well-being, problems, risk, and functioning. Items are scored on a scale from 0 (never) to 4 (always or almost always). Higher scores indicate greater psychological distress. This instrument is suitable as an initial assessment tool and as an outcome measure. The Spanish versionof this measure will be used. This version was translated by Feixas et al. (2012) and has shown good psychometric properties in Spain (Trujillo et al. 2016) and Ecuador (Paz et al. 2020).
Change in Clinical Outcomes in Routine Evaluation-10 (CORE-10) | CORE-10 is administered to adult clients at the second week and then routinely every week until treatment completion
  The CORE-10 (Barkham et al., 2013) is a generic, short, and easy-to-use assessment measure. Its items were drawn from the CORE-OM. The CORE-10 is an instrument that has shown good psychometric properties (Barkham et al., 2013) and is practical for use on a session-by-session basis with people presenting with psychological distress in mental health settings. Its Spanish version will be used (Feixas et al., 2012).
Change in Young Person's-Clinical Outcomes in Routine Evaluation (YP-CORE) | YP-CORE is administered to adolescent clients at baseline and then routinely every week until treatment completion
  The YP-CORE is a brief self-report instrument capable of detecting psychological distress in adolescents, generated by a wide range of problems, while providing information about the person's general functioning (Twigg et al., 2009). It has 10 items, which must be answered on a 5-point scale (0 to 4). Its Spanish version will be used. The YP-CORE was translated to Spanish by Feixas et al. (2018) and showed adequate psychometric properties. In the present study, we will use a version of this measure adapted for Ecuador and Latin America whose psychometric properties are being explored.

SECONDARY OUTCOMES:
Change in Life Satisfaction Scale | Life Satisfaction Scale is administered to all clients at baseline and immediately after treatment completion
  It is a 10-point scale that asks respondents to rate their degree of satisfaction with life in the present. It will be presented in Spanish.
Change in Ambivalence in Psychotherapy Questionnaire (APQ) | APQ is administered to adult clients at baseline and then routinely every four weeks
  It is a 9-item scale that measures the level of ambivalence towards change perceived by the consultants. It includes two subscales, demoralization and oscillation, and an overall score of ambivalence towards change (Oliveira et al., 2020). Both the original version (Oliveira et al., 2020) and the Spanish version (Montesano et al., submitted for publication) have demonstrated good psychometric properties, including good convergent and divergent validity. In this study the Spanish version will be used.
Change in Systemic Clinical Outcome and Routine Evaluation-15 (SCORE-15) | SCORE-15 is administered to all clients at baseline, at four weeks and immediately after treatment completion
  It is a 15-item questionnaire with a scale of 1 to 5, where 1 means "strongly disagree" and 5 means "strongly agree". It was designed to be completed by family members, aged 12 years or older (Stratton et al., 2010). It has three dimensions: strengths, difficulties and communication. Lower scores correspond to better family functioning. In addition, the SCORE-15 has two scales ranging from 1 to 10 on which participants rate the perceived effectiveness of the therapeutic intervention and the perceived severity of the difficulty leading to treatment. In the present study, we will use the Spanish version of this measure which has shown adequate reliability and validity in a Spanish sample (Rivas & Pereira, 2016).
Satisfaction with the Treatment Received Scale (CRES-4) | CRES-4 is administered to all clients immediately after treatment completion
  The CRES-4 scale has 4 items: one question on satisfaction, one on the level of resolution of the main problem, one on the emotional state before the start of treatment and one question on the emotional state when completing the questionnaire (Feixas et al., 2012). These questions allow interpretations to be made about the perceived change in their emotional state, satisfaction and resolution of the problem. In this study, the Spanish version of this measure will be used (Feixas et al., 2012).
Change in Therapeutic Alliance Scale | Therapeutic Alliance Scale is administered to all clients immediately after the first intervention and then routinely every week until treatment completion
  It is a 10-point one-item measure that evaluates therapeutic alliance. Clients are asked to state, in general, how connected they feel to their therapist and if they have talked about what the clients were interested in addressing in therapy. It will be presented in Spanish.

OTHER OUTCOMES:
CORE Therapy Assessment Form (TAF) | CORE TAF is completed at baseline
  The CORE TAF is a pragmatic form designed to be filled out by therapists at baseline. The CORE-TAF includes referral information, sociodemographic data on the client, and data on the nature, severity, and duration of the client's problems. (Barkham et al., 2015; Evans 2003). We will use its Spanish version, which is currently being translated.
CORE End of Therapy (EoT) | CORE EoT is completed immediately after treatment completion
  The CORE EoT is a pragmatic form designed to be filled out by therapists immediately after treatment completion. The CORE-EoT reports on the completed treatment, including the number of sessions, type of therapy, length and frequency of sessions, whether the ending was planned or unplanned, and the potential benefits of therapy (Barkham et al., 2015; Evans 2003). We will use its Spanish version, which is currently being translated.

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Valdiviezo-Oña, MSc, Principal Investigator — University of Americas; Clara Paz, PhD, Study Director — University of Americas; Adrián Montesano del Campo, PhD, Study Director — Universitat Oberta de Catalunya
Locations (1):
- Centro de Psicología Aplicada, Quito, Pichincha, Ecuador

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Barkham M, Bewick B, Mullin T, Gilbody S, Connell J, Cahill J, Mellor-Clark J, Richards D, Unsworth G, Evans C. The CORE-10: A short measure of psychological distress for routine use in the psychological therapies. Counselling and Psychotherapy Research. 2013; 13(1): 3-13.
- [Background] Barkham M, Mellor-Clark J, Stiles WB. A CORE approach to progress monitoring and feedback: Enhancing evidence and improving practice. Psychotherapy (Chic). 2015 Dec;52(4):402-11. doi: 10.1037/pst0000030. PMID 26641370
- [Background] Evans C, Connell J, Barkham M, Margison F, McGrath G, Mellor-Clark J, Audin K. Towards a standardised brief outcome measure: psychometric properties and utility of the CORE-OM. Br J Psychiatry. 2002 Jan;180:51-60. doi: 10.1192/bjp.180.1.51. PMID 11772852
- [Background] Evans C, Connell J, Barkham M, Marshall C, Mellor-Clark J. Practice-based evidence: benchmarking NHS primary care counselling services at national and local levels. Clinical Psychology & Psychotherapy: An International Journal of Theory & Practice. 2003; 10(6): 374-388
- [Background] Feixas G, Badia E, Bados A, Medina JC, Grau A, Magallon E, Botella L, Evans C. Adaptation and psychometric properties of the spanish version of the yp-core (Young Person's Clinical Outcomes in Routine Evaluation). Actas Esp Psiquiatr. 2018 May;46(3):75-82. Epub 2018 May 1. PMID 29892966
- [Background] Feixas G, Evans C, Trujillo A, Saúl LÁ, Botella L, Corbella S, González S, Bados A, Garcia-Grau A, López-González. M. La version española del CORE-OM: Clinical Outcomes in Routine Evaluation - Outcome Measure. Revista de Psicoterapia. 2012; 23(89): 109-135.
- [Background] Feixas, G, Pucurull O, Roca C, Paz C, García-Grau E, Bados, A. Escala de satisfacción con el tratamiento recibido (CRES-4): la versión en español. Revista de Psicoterapia. 2012; 23(89): 51-58.
- [Background] Oliveira JT, Ribeiro AP, Goncalves MM. Ambivalence in Psychotherapy Questionnaire: Development and validation studies. Clin Psychol Psychother. 2020 Sep;27(5):727-735. doi: 10.1002/cpp.2457. Epub 2020 Apr 27. PMID 32285558
- [Background] Paz C, Mascialino G, Evans C. Exploration of the psychometric properties of the Clinical Outcomes in Routine Evaluation-Outcome Measure in Ecuador. BMC Psychol. 2020 Sep 1;8(1):94. doi: 10.1186/s40359-020-00443-z. PMID 32873334
- [Background] Rivas G, Pereira R. Validación de una escala de evaluación familiar: adaptación del SCORE-15 con normas en español. Mosaico: revista de la Federación Española de Asociaciones de Terapia Familiar. 2016; 63: 16-28.
- [Background] Stratton P, Bland J, Janes E, Lask J. Developing an indicator of family function and a practicable outcome measure for systemic family and couple therapy: the SCORE. Journal of family therapy. 2010; 32(3): 232-258.
- [Background] Trujillo A, Feixas G, Bados A, Garcia-Grau E, Salla M, Medina JC, Montesano A, Soriano J, Medeiros-Ferreira L, Canete J, Corbella S, Grau A, Lana F, Evans C. Psychometric properties of the Spanish version of the Clinical Outcomes in Routine Evaluation - Outcome Measure. Neuropsychiatr Dis Treat. 2016 Jun 21;12:1457-66. doi: 10.2147/NDT.S103079. eCollection 2016. PMID 27382288
- [Background] Twigg E, Barkham M, Bewick BM, Mulhern B, Connell J, Cooper M. The YP-CORE: Development and validation of a young person's version of the CORE-OM. Counselling and Psychotherapy Research. 2009; 9: 160-168.
- [Derived] Valdiviezo-Ona J, Montesano A, Evans C, Paz C. Fostering practice-based evidence through routine outcome monitoring in a university psychotherapy service for common mental health problems: a protocol for a naturalistic, observational study. BMJ Open. 2023 May 24;13(5):e071875. doi: 10.1136/bmjopen-2023-071875. PMID 37225267